CLINICAL TRIAL: NCT05439785
Title: A Comparison of Plaque Control Efficacy Between Interdental Brushes Versus Dental Floss in Patients With Periodontal Disease
Brief Title: Plaque Control Efficacy Between Interdental Brushes Versus Dental Floss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Dental College (Other)
Responsible Party: Principal Investigator, Madiha Sultan, Principal Investigator, Post Graduate Trainee Specialty of Periodontology,, Fatima Jinnah Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FatimaJDC420
Record Dates: First submitted 2022-06-06; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Periodontal Diseases; Dental Plaque
MeSH Terms: conditions — Periodontal Diseases; Dental Plaque | interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Dental floss
  Interventions: Device: Dental floss/Interdental brush
- Group 2 (Experimental): Interdental brush
  Interventions: Device: Dental floss/Interdental brush

INTERVENTIONS:
Device: Dental floss/Interdental brush — Initially plaque disclosing tablets were used to disclose plaque and plaque and bleeding scores will be recoded. After mechanical plaque debrided, instructions regarding the allocated interdental device given to the patient along with motivation to continue practicing good oral hygiene. After six weeks patients were recalled for reevaluation

SUMMARY:
The purpose of this study is to compare between plaque control efficacy of interdental brushes versus interdental floss , for the prevention of periodontal disease (gingivitis) and to determine the most convenient routine interdental plaque control method amongst the two

ELIGIBILITY:
Inclusion Criteria:

* All patients above 18 years of age with gingivitis
* patients of both gender

Exclusion Criteria:

* patients who refuse participate in the study
* patients with systemic medical problems
* patients using medications that may affect gingival tissue (overgrowth/bleeding)
* patients habitual of betel nut/tobacco smoking/substance abuse
* patients with fluorosis or any other enamel and dentinal deformity
* pregnant women
* patients undergoing orthodontic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plaque score records according to Silness and Loe and O'Leary et al plaque score/index at week 6 | baseline and week 6
  Silness and Loe Plaque Index and O'Leary et al plaque index are used as tools to measure plaque score by disclosing plaque, using a chewable plaque disclosing tablet. Possible score range from 0 (absence of microbial plaque) to 3 (large amount of plaque in sulcus or pocket along the free gingiva margin). Change = ( week 6 score - baseline score)

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Jinnah Dental College and Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No